CLINICAL TRIAL: NCT06824454
Title: Evaluation of Dipyridamole in Preventing Post-Transplant Hypophosphatemia in Kidney Transplant Recipients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephan Busque, Professor of Surgery (Abdominal Transplantation), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76830
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Hypophosphatemia; Kidney Transplantation
Keywords: Post-kidney transplant care; Dipyridamole; Renal phosphate loss; Serum phosphate levels; Phosphate supplementation; Transplant graft function; Kidney transplant complications
MeSH Terms: conditions — Hypophosphatemia | interventions — Dipyridamole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Participants receive Dipyridamole in addition to standard post-transplant care.
  Interventions: Drug: Dipyridamole 75 MG
- Control Group (No Intervention): Participants in this group will receive standard post-transplant care without Dipyridamole.

INTERVENTIONS:
Drug: Dipyridamole 75 MG — Dipyridamole administered three times daily when serum phosphorus levels fall below 4 mg/dL. The drug is used off-label for this study to manage hypophosphatemia in kidney transplant recipients.
  Arms: Treatment Group

SUMMARY:
The primary goal is to determine if Dipyridamole can improve serum phosphate levels and reduce the need for phosphate supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant patients.
* No known contraindications to Dipyridamole

Exclusion Criteria:

* Contraindications to Dipyridamole.
* Patients with delayed graft function (defined as the need for dialysis within seven days post-transplantation).
* Patients requiring Plavix, direct oral anticoagulants (DOACs), or Coumadin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Phosphorus Levels After Dipyridamole Administration | Baseline, 1 week, 4 weeks, 8 weeks, 12 weeks, and after stopping medicatio
  This study will evaluate the effectiveness of Dipyridamole in increasing serum phosphorus levels in kidney transplant recipients with hypophosphatemia.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Busque, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No